CLINICAL TRIAL: NCT05018078
Title: The Fifth Medical Center of Chinese PLA General Hospital
Brief Title: Safety and Immunogenicity of COVID-19 Vaccination in Patients With Cancer
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ky-2021-7-9-1
Record Dates: First submitted 2021-08-18; First posted 2021-08-24 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Patients With Cancers; COVID-19; Vaccine
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Coronavirus vaccination (Experimental): Patients in the experimental need to accept the coronavirus vaccination
  Interventions: Biological: Coronavirus vaccine

INTERVENTIONS:
Biological: Coronavirus vaccine — Coronavirus vaccine was inoculated on day 0 and day 25±3, respectively

SUMMARY:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) has caused pandemic since outbreak in 2020. Patients with cancers may be at higher risk than those without cancer for coronavirus disease 2019 (COVID-19). At present, limited data are available on the safety and immunogenicity of COVID-19 vaccination for patients with cancer.

DETAILED DESCRIPTION:
This study is a prospective, single-arm, open-label clinical trial. A total of 300 patients with different cancers including hepatocellular carcinoma, breast cancer, lung cancer, esophageal cancer, gastric cancer and colorectal cancer were included in this vaccination study. All of the patients will further accept 12 months follow-up study after vaccination. Safety and immunogenicity will be carefully recorded and detected.

ELIGIBILITY:
Inclusion Criteria:

1. Age above 18 years
2. Patients with diagnosed cancers including hepatocellular carcinoma, breast cancer, lung cancer, esophageal cancer, gastric cancer and colorectal cancer were included .
3. Patients who have received local or systemic anti-cancer therapies according to the treatment guidelines previously or currently, and have a stable condition with the ECOG score below 2.
4. The functions of multi-organs were normal or basically normal, and there are no contraindications for vaccination.

Exclusion Criteria:

1. Patients with acute attack of chronic diseases.
2. Patients have history of convulsion, epilepsy, encephalopathy and psychosis.
3. Patients who are allergic to any component of the vaccine, or have a serious history of vaccine allergy.
4. Pregnant or lactating women.
5. Sufferring serious cardiovascular diseases, such as arrhythmia, conduction block, myocardial infarction, and severe hypertension can not be well controlled by drugs.
6. Patients have severe chronic diseases or diseases can not be controlled well during the progress, such as asthma, diabetes, thyroid disease, etc. Congenital or acquired angioedema / neuroedema.
7. Systemic cytotoxic drugs, cell therapies including NK cells, cytokine induced killer cells, Dendritic cells, CTL and stem cells infusion are required during vaccination.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2021-08-30 (Actual); Primary Completion 2023-08-30 (Estimated); Study Completion 2023-10-30 (Estimated)

PRIMARY OUTCOMES:
Safety of coronavirus vaccine | Within 2 months after the first dose of coronavirus vaccine
  Occurence of adverse effects after COVID-19 vaccination
Immunogenicity of coronavirus vaccine | Within 2 months after the first dose of coronavirus vaccine
  Titers of anti-SARS-CoV-2 antibodies

SECONDARY OUTCOMES:
Safety of coronavirus vaccine | Within 13 months after the first dose of coronavirus vaccine
  Occurence of adverse effects after COVID-19 vaccination
Immunogenicity of coronavirus vaccine | Within 13 months after the first dose of coronavirus vaccine
  Titers of anti-SARS-CoV-2 antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Shu-juan Li, MD, Study Director — Beijing 302 Hospital
Locations (1):
- The Fifth Medical Center of PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lai CC, Wang JH, Hsueh PR. Population-based seroprevalence surveys of anti-SARS-CoV-2 antibody: An up-to-date review. Int J Infect Dis. 2020 Dec;101:314-322. doi: 10.1016/j.ijid.2020.10.011. Epub 2020 Oct 9. PMID 33045429
- [Background] Dai M, Liu D, Liu M, Zhou F, Li G, Chen Z, Zhang Z, You H, Wu M, Zheng Q, Xiong Y, Xiong H, Wang C, Chen C, Xiong F, Zhang Y, Peng Y, Ge S, Zhen B, Yu T, Wang L, Wang H, Liu Y, Chen Y, Mei J, Gao X, Li Z, Gan L, He C, Li Z, Shi Y, Qi Y, Yang J, Tenen DG, Chai L, Mucci LA, Santillana M, Cai H. Patients with Cancer Appear More Vulnerable to SARS-CoV-2: A Multicenter Study during the COVID-19 Outbreak. Cancer Discov. 2020 Jun;10(6):783-791. doi: 10.1158/2159-8290.CD-20-0422. Epub 2020 Apr 28. PMID 32345594
- [Background] Monin L, Laing AG, Munoz-Ruiz M, McKenzie DR, Del Molino Del Barrio I, Alaguthurai T, Domingo-Vila C, Hayday TS, Graham C, Seow J, Abdul-Jawad S, Kamdar S, Harvey-Jones E, Graham R, Cooper J, Khan M, Vidler J, Kakkassery H, Sinha S, Davis R, Dupont L, Francos Quijorna I, O'Brien-Gore C, Lee PL, Eum J, Conde Poole M, Joseph M, Davies D, Wu Y, Swampillai A, North BV, Montes A, Harries M, Rigg A, Spicer J, Malim MH, Fields P, Patten P, Di Rosa F, Papa S, Tree T, Doores KJ, Hayday AC, Irshad S. Safety and immunogenicity of one versus two doses of the COVID-19 vaccine BNT162b2 for patients with cancer: interim analysis of a prospective observational study. Lancet Oncol. 2021 Jun;22(6):765-778. doi: 10.1016/S1470-2045(21)00213-8. Epub 2021 Apr 27. PMID 33930323
- [Background] Herishanu Y, Avivi I, Aharon A, Shefer G, Levi S, Bronstein Y, Morales M, Ziv T, Shorer Arbel Y, Scarfo L, Joffe E, Perry C, Ghia P. Efficacy of the BNT162b2 mRNA COVID-19 vaccine in patients with chronic lymphocytic leukemia. Blood. 2021 Jun 10;137(23):3165-3173. doi: 10.1182/blood.2021011568. PMID 33861303
- [Background] Cornberg M, Buti M, Eberhardt CS, Grossi PA, Shouval D. EASL position paper on the use of COVID-19 vaccines in patients with chronic liver diseases, hepatobiliary cancer and liver transplant recipients. J Hepatol. 2021 Apr;74(4):944-951. doi: 10.1016/j.jhep.2021.01.032. Epub 2021 Feb 6. PMID 33563499
- [Background] Fix OK, Blumberg EA, Chang KM, Chu J, Chung RT, Goacher EK, Hameed B, Kaul DR, Kulik LM, Kwok RM, McGuire BM, Mulligan DC, Price JC, Reau NS, Reddy KR, Reynolds A, Rosen HR, Russo MW, Schilsky ML, Verna EC, Ward JW, Fontana RJ; AASLD COVID-19 Vaccine Working Group. American Association for the Study of Liver Diseases Expert Panel Consensus Statement: Vaccines to Prevent Coronavirus Disease 2019 Infection in Patients With Liver Disease. Hepatology. 2021 Aug;74(2):1049-1064. doi: 10.1002/hep.31751. PMID 33577086